CLINICAL TRIAL: NCT03143335
Title: Direct to Implant Extracellular Matrix Hammock Based pre-or Retropectoral Breast Reconstruction
Brief Title: Direct to Implant Breast Reconstruction Based Pre- or Retropectoral
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Odense University Hospital (Other)
Collaborators: Sygehus Lillebaelt (Other); Sykehuset Telemark (Other Government)
Responsible Party: Principal Investigator, Diana Lydia Dyrberg, Medical Doctor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-2016060
Record Dates: First submitted 2017-05-01; First posted 2017-05-08 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Breast Reconstruction
Keywords: Breast; Reconstruction; BAD; Implant; ADM

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retropectoral immediate breast reconstruction (Active Comparator): Participants are randomized to immediate breast reconstruction with the implant placed retropectoral.
  Interventions: Procedure: Retropectoral immediate breast reconstruction
- Prepectoral immediate breast reconstruction (Active Comparator): Participants are randomized to direct to immediate breast reconstruction with the implant placed prepectoral using acellular dermal matrix for support.
  Interventions: Procedure: Prepectoral immediate breast reconstruction

INTERVENTIONS:
Procedure: Retropectoral immediate breast reconstruction — Immediate reconstruction with the implant placed in a standard fashion, i.e. retropectoral in combination with an acellular dermal matrix.
  Arms: Retropectoral immediate breast reconstruction
Procedure: Prepectoral immediate breast reconstruction — Immediate breast reconstruction with the implant placed prepectoral supported by acellular dermal matrix alone.
  Arms: Prepectoral immediate breast reconstruction

SUMMARY:
The purpose of this study is to examine different outcomes of breast reconstruction in women who are treated for breast cancer with skin sparing mastectomy and subsequently a primary implant based reconstruction by one of two different techniques with either a pre- or retropectoral placement of the implant.

The main objective of the study is to establish whether one of these techniques may result in a superior outcome and thus should be recommended as first choice treatment rather than the other.

DETAILED DESCRIPTION:
Women diagnosed with breast cancer, large areas of ductal carcinoma in situ or a hereditary high risk of breast cancer are offered a mastectomy either as a therapeutic or a risk reducing intervention. Those, who are found eligible for an immediate breast reconstruction using an implant are reconstructed by either a skin sparing mastectomy (SSM) or a nipple sparing mastectomy (NSM) using an extracellular matrix. The current technique is to place the implant in a retropectoral pocket in which the cranial part of the implant is covered by the major pectoral muscle, whereas the caudal part of the implant is covered and supported by an extracellular dermal matrix (ADM) as a hammock.

Recent focus on the functional outcome has, however, identified a new challenge - breast animation deformity (BAD), breast distortion or "jumping breast". The consequence of the condition is that women with aesthetic pleasant results, in rest, experience breast animation deformity during contraction of the major pectoral muscle. Evaluation of forty breast augmented women with a subpectoral positioning of the implant revealed that 77.5% had some kind of distortion during movement of the arm. In these healthy individuals, however, the condition is partly hidden by the glandular tissue and subcutaneous fatty tissue.

The condition is more severe in women with a reconstructed breast using a retropectorally placed implant, where the glandular tissue has been removed, leaving only the subcutaneous fatty tissue to cover the muscle and implant. The investigators know from experience and from reviewing unpublished clinical pictures and videos of thirty patients, who had an immediate breast reconstruction using the hammock technique, that the vast majority of patients have a pronounced degree of BAD.

Patients, who have a prepectoral placement of their implant, tend to have a lesser degree of BAD. The functional outcome of the prepectoral placement of the implant has previously not been compared to the retropectoral placement of the implant in women reconstructed by an implant and an ADM. A possible disadvantage of a prepectoral placement of the implant may be less soft-tissue coverage supplied by the pectoral muscle leading to higher risk of significant capsular formation. Less soft-tissue coverage may also result in a more visible implant border and rippling. Furthermore, the implant will not benefit from the abundant vascularity of the muscle and in theory perhaps not be as resistant to infections and implant loss as the subpectoral positioned implants.

The primary aim of this study is to compare the degree of BAD following a prepectoral to a retropectoral placement of the implant using the hammock for immediate breast reconstruction. For this purpose we have designed two separate trials:

Retrospective Follow-up trial: The investigators plan to invite a total of forty patients to compare breast animation deformity and shoulder and arm morbidity in a retrospective cohort of patients. Twenty patients, who have had a conventional immediate breast reconstruction with a retropectoral placement of the implant will be compared to twenty patients , who have had an immediate breast reconstruction with a prepectoral placement of the implant.

Randomized clinical trial: Investigators plan to collect, examine and compare data on the two surgical techniques in order to test superiority of the prepectoral implant based reconstruction in accordance with our hypothesis that it leads to lesser degree of BAD and better functional outcomes.

The trial is thus designed with two parallel study-arms as participants are allocated to reconstruction by either retro- or prepectoral placement of the implant in the ratio 1:1.

As the clinically most important parameter seems to be breast animation deformity this will serve as primary end-point. Functional changes in shoulder and arm function between the two surgical techniques is also a very important perimeter to investigate and will be analysed as secondary end-points.

In addition to the above data a number of other patient related outcomes will be collected as part of this trial.

Designed as a multicentre trial, participant enrollment and data Collection will be performed at academic Hospitals in Denmark and Norway.

A password protected Electronic database placed on a secure server will be established. This database will only be accessible to the primary investigator of the research Group who will be involved in the analysis of the data.

This study will provide a better knowledge of the expected outcome of immediate breast reconstruction, when it is performed by one of these two surgical techniques. The investigators expect that these results will help determine if the prepectoral implant placement may represent a better and gentler method for reconstruction of the breast with lower morbidity than the retropectoral implant placement. In all cases the results of this trial will enable us to provide our patients with better and more objective information, before they are subjected to immediate breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

Women over 18 years referred to the Department of plastic surgery, Odense University Hospital, Lillebaelt Hospital Vejle, Denmark or Telemark Hospital, Skien, Norway between January 2017 and July 2018, who are found eligible for immediate breast reconstruction.

Exclusion Criteria:

1. Dementia that makes it impossible to obtain informed consent
2. Non-Danish speaking patients from whom informed consent cannot be obtained by interpreter
3. Tobacco users
4. Women with known hypertension treated with more than one drug
5. Women who had pre-surgical radiation therapy.
6. Women planned to have postsurgical radiation therapy.
7. BMI above 32 or below 22

However, the final decision relies on sufficient thickness of the skin flaps after mastectomy prior to immediate reconstruction.

Invited patient will receive both oral and written participant information after which there will be as many days for reflection as the treatment guaranty for cancer allows.

Patients considering participation will be invited for a second consultation where written informed consent will be obtained from all who accept the invitation. Randomization will be performed during surgery, prior to reconstruction. Patients who do not wish to participate will be reconstruction with the implant placed retropectoral.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Breast animation deformity | 12 months
  Breast animation deformity (BAD) is one of the more unpleasant cosmetic results that can be seen after breast reconstruction with a retropectoral placed implant. The degree of breast distortion will be evaluated by two experienced plastic surgeons and classified according to the published classification by Spear S. Because the degree of breast distortion will be the primary outcome measure of this randomised trial, the sample size will be based on assumptions regarding the grade of distortion between groups. For this purpose, the distortion will be divided into two groups: 1) Severe distortion containing degree 3 and 4 and 2) Moderate distortion containing degree 1 and 2. In bilateral cases the most severe side will be the one used for comparison

SECONDARY OUTCOMES:
Shoulder function | 3 and 12 months
  Because one of the most important difference between the two surgical procedures is the involvement of the major pectoralis muscle, change in shoulder function is relevant to investigate. For evaluation investigators use the internationally validated Constant Shoulder Score (CSS). This system assess pain, function in everyday life, range of motion and strength and incorporates these parameters into one total score. It is the recommended scoring-system by the European Society of Shoulder and Elbow Surgery. Each variable in the system is evaluated separately. For all participants scoring will be performed preoperatively as well as 3 and 12 months postoperatively. Shoulder function will be evaluated bilaterally at all stages. To avoid multiplicity-issues the primary end point has been defined as the difference in total score between the baseline evaluation preoperatively and the evaluation one year postoperatively.

OTHER OUTCOMES:
Quality of Life | 12 months
  The participants quality of life will be assessed before and after reconstruction using the international validated questionnaire BREAST-Q.
Postoperative pain | 3 months
  Investigators believe that the pectoralis muscle involvement is responsible for much of the postoperative pain and wish to test this theory by monitoring on a pain scale (VAS) from 0-10. This will be monitored on regular hours post operatively and the use of postoperative analgesics will be rated.
Postoperative complications | 3 months
  Complications following immediate breast reconstruction have been described in numerous papers. Investigators will record skin necrosis, wound dehiscence, infection, seromas, bleeding and explantation of the implant. Complications will be classified as either major or minor depending on the need for surgical revision in general anaesthesia. Complication rates will be compared between the two groups.
Fat-grafting and surgical corrections | 12 months
  In order to improve the cosmetic and functional result of breast reconstruction participants in this study will be treated by fatgrafting when needed. The number of post-reconstructive fatgrafting and surgical corrections within the first 12 months will be recorded.
Length of stay | 1 month
  In order to evaluate if there is a difference in inpatient days between each surgical technique investigators record duration of hospitalization and days until removal of the drains for all participants.
Capsular contraction | 12 months
  After 12 months all participants will be evaluated and examined by two experienced plastic surgeons where the grade of capsular contraction will evaluated by Bakers classification.
Aesthetic result | 12 months
  All participants will be asked to evaluate the appearance of their breasts on a scale from to 10 before surgery and once again 12 months after surgery. Furthermore, participants will have their breast photographed by a professional photographer and video recordings will also be obtained. Video recordings and photographs will be evaluated by two unbiased consultant plastic surgeons that aren't associated with neither the department nor the project. These specialists will perform the same evaluation as the participants, as these results will be compared to the participants´ own perception. Furthermore, the two consultant plastic surgeons will be asked to evaluate specific parameters as rippling and visibility of implant borders cranially and classify them as either optimum, good, borderline or poor. Based on this we will conduct an inter observer reliability test.
Temperature evaluation | 3 and 12 months
  All participating patients will be asked if they experience the reconstructed breast colder than previous after 3 and 12 months to see if there is a significant difference in sensation of "Coldness" of the breast.

CONTACTS AND LOCATIONS:
Overall Officials: Jørn Bo JB Thomsen, MD, PhD, Study Chair — Center Hospital Vejle, Institute of Regional Health Research, University of Southern Denmark
Locations (3):
- Denmark (2):
  - Odense University Hospital, Odense
  - Lillebaelt Hospital Vejle, Vejle
- Telemark Hospital, Skien, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dyrberg DL, Gunnarsson GL, Bille C, Sorensen JA, Thomsen JB. Direct-to-Implant Extracellular Matrix Hammock-based Breast Reconstruction; Prepectoral or Subpectoral? Trials. 2020 Feb 10;21(1):160. doi: 10.1186/s13063-020-4125-6. PMID 32041661